CLINICAL TRIAL: NCT05298527
Title: THE EFFECT OF BACK MASSAGE APPLIED BY PARTNERS TO CLIMACTERIC WOMEN WITH SLEEP PROBLEM ON MENOPAUSAL COMPLAINTS, SLEEP QUALITY AND MARITAL ADJUSTMENT
Brief Title: BACK MASSAGE APPLIED CLIMACTERIC WOMEN MENOPAUSAL COMPLAINTS, SLEEP QUALITY AND MARITAL ADJUSTMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, DİDEM KAYA, Assistant Professor Doctor, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NuhNaciYazganU
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Climactericum; Sleep
Keywords: climacteric period; menopausal complaint; back massage; sleep quality; marital adjustment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study was conducted as the randomized controlled experimental trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In this study, the purpose of the study was explained to the women from intervention group and their partners by visiting them in their home. Personal Information Form (PIF), Pittsburgh Sleep Quality Index (PSQI), Menopause Symptoms Rating Scale (MSRS) and Marital Adjustment Scale (MAS) were filled by the women and MAS was filled by their partners. Firstly, back massage was taught to the partners of women in the intervention group. The massage was made half an hour before the women's sleep time for a total of 15 minutes. Partners were ensured to apply this massage twice a week for four weeks. The intervention group was called by telephone every week to ensure continuity of the study. By visiting those at their homes again at the end of the fourth week, PSQI, MSRS, and MAS were filled by the women and MAS was filled by their husbands for the last time.
  Interventions: Behavioral: Back Massage
- Control Group (No Intervention): In this study, the purpose of the study was explained to the women from control group and their partners by visiting them in their home. Their signatures indicating that they agreed to participate in the study were obtained after having them read the informed consent form. Personal Information Form (PIF), Pittsburgh Sleep Quality Index (PSQI), Menopause Symptoms Rating Scale (MSRS) and Marital Adjustment Scale (MAS) were filled by the women and MAS was filled by their partners. No application was made to the couples in the control group. By visiting those at their homes again at the end of the fourth week, PSQI, MSRS, and MAS were filled by the women and MAS was filled by their husbands for the last time. Back massage training was given to the partners of the women in the control group at the end of the fourth week.

INTERVENTIONS:
Behavioral: Back Massage — The woman lies face down and a pillow is placed under her forehead. Massage begins with effleurage. Petrissage is started from the sacrum and the hands are lifted up to the nape and repeated 4 times. After the petrissage movement is completed, effusion is applied to the area once. Friction is applied. After rubbing, tapotement is applied to the entire back.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine the effect of back massage applied by partners on menopausal complaints, sleep quality, and marital adjustment of women in climacteric period.

DETAILED DESCRIPTION:
Climacterium is a life period in which women move from the reproductive age to the period when their reproductive ability is lost due to the decrease in ovarian functions. The most common climacteric disorder is vasomotor changes. The most common problem seen in menopausal period after vasomotor complaints is insomnia.

Sleep disorders seen in climacteric period negatively affect the quality of life and psychosocial health of woman. In their study, Jean-Louis et al., expressed that women in menopausal period spent approximately 10% of their daily sleep time by sleeping outside the bed during the day. 61% of menopausal women woke up at least once a week and several times from the night's sleep. In their study, Anttalainen et al., determined that women in postmenopausal period had more sleep problems compared to women in premenopausal period. In addition to physical changes due to hormonal changes in climacterium, mental problems such as nervousness, anxiety and depression developing in women may negatively affect the relationships in family environment especially the communication with the spouse. Besides, it is thought that an incompatible marriage can increase menopausal complaints. In the studies investigating the relationship between menopausal complaints and marital adjustment, women with compatible marital life were found to experience less menopausal complaints. Due to the negative effects of physician-controlled hormone replacement treatment administered to reduce menopausal symptoms, demand for non-pharmacological interventions has increased and women have started to accept that therapeutic massage is safe and contributes to health. It is stated that women experience insomnia, a symptom of menopause, and tend to choose especially body therapies from alternative therapies in the first place. Massage is widely accepted as a treatment tool. Although the menopausal period is physiological, it is a period that must be addressed specifically by healthcare professionals since it is accompanied by pathological events causing distress in life and impairing the quality of life.

The purpose of this study is to determine the effect of back massage applied by partners on menopausal complaints, sleep quality, and marital adjustment of women in climacteric period.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 40-65 years,
* women who have 5 or more points from Pittsburgh Sleep Quality Index (PSQI),
* women who do not use hormone therapy or who stopped hormone therapy at least one year ago.

Exclusion Criteria:

* women who had sleep problems before climacteric period,
* women who had uncontrolled chronic disease,
* women receiving psychiatric treatment and/or using sleeping pills,
* women with open wounds on their back were excluded from the study group.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 4 minutes
  It is a scale developed by Buysse et al., in 1989. Its validity and reliability study was conducted in 1996 by Ağargün et al. PSQI provides a quantitative measure of sleep quality. There are 24 questions in the scale and 19 of these questions are self-rated. PSQI total score of 5 or higher indicates poor sleep quality. The Cronbach's alpha internal consistency coefficient of the scale, whose validity and reliability was conducted by Ağargün et al. was determined as 0.80.
Menopause Symptoms Rating Scale (MSRS) | 2 minutes
  The Menopause Symptoms Rating Scale, originally called as Menopause Rating Scale, was developed in German by Schneider, Heinemann et al. in 1992 to determine the severity of menopausal symptoms and their effect on quality of life. The English adaptation, validity and reliability of the scale were conducted in 1996 by Schneider, Heinemann et al. The validity and reliability study of the scale was conducted in Turkey by Özlem Can Gürkan. The minimum score of the scale is "0" and the maximum score is "44". The high total score of the scale indicates that both quality of life is low and menopausal complaints are high. In the validity and reliability study by Gürkan, the Cronbach's alpha internal consistency coefficient was found as 0.84.
Marital Adjustment Scale (MAS) | 3 minutes
  MAS, developed by Locke and Wallace in 1959, is composed of 15 items. The validity and reliability of the scale was conducted by Tutarel-Kışlak in 1999. It was found that the scale can significantly distinguish coupes with and without marital problems. The cut-off point of the scale is 43. While scores lower than 43 refer to a general marital maladjustment, scores higher than 43 indicate overall marital adjustment. In the validity and reliability study of Tutarel-Kışlak, the Cronbach's alpha internal consistency coefficient of the scale was found as 0.90.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Kocasinan/Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Jean-Louis G, Kripke DF, Assmus JD, Langer RD. Sleep-wake patterns among postmenopausal women: a 24-hour unattended polysomnographic study. J Gerontol A Biol Sci Med Sci. 2000 Mar;55(3):M120-3. doi: 10.1093/gerona/55.3.m120. PMID 10795722
- [Background] Kripke DF, Brunner R, Freeman R, Hendrix SL, Jackson RD, Masaki K, Carter RA. Sleep Complaints of Postmenopausal Women. Clin J Womens Health. 2001 Dec 1;1(5):244-252. doi: 10.1053/cjwh.2001.30491. PMID 21461131
- [Background] Anttalainen U, Saaresranta T, Aittokallio J, Kalleinen N, Vahlberg T, Virtanen I, Polo O. Impact of menopause on the manifestation and severity of sleep-disordered breathing. Acta Obstet Gynecol Scand. 2006;85(11):1381-8. doi: 10.1080/00016340600935649. PMID 17091421
- [Background] Hachul H, Oliveira DS, Bittencourt LR, Andersen ML, Tufik S. The beneficial effects of massage therapy for insomnia in postmenopausal women. Sleep Sci. 2014 Jun;7(2):114-6. doi: 10.1016/j.slsci.2014.09.005. Epub 2014 Sep 16. PMID 26483913
- [Background] Newton KM, Buist DS, Keenan NL, Anderson LA, LaCroix AZ. Use of alternative therapies for menopause symptoms: results of a population-based survey. Obstet Gynecol. 2002 Jul;100(1):18-25. doi: 10.1016/s0029-7844(02)02005-7. PMID 12100799
- [Background] Oliveira D, Hachul H, Tufik S, Bittencourt L. Effect of massage in postmenopausal women with insomnia: a pilot study. Clinics (Sao Paulo). 2011;66(2):343-6. doi: 10.1590/s1807-59322011000200026. No abstract available. PMID 21484056
- [Background] Oliveira DS, Hachul H, Goto V, Tufik S, Bittencourt LR. Effect of therapeutic massage on insomnia and climacteric symptoms in postmenopausal women. Climacteric. 2012 Feb;15(1):21-9. doi: 10.3109/13697137.2011.587557. Epub 2011 Oct 23. PMID 22017318